CLINICAL TRIAL: NCT03330847
Title: A Phase II, Open Label, Randomised, Multi-centre Study to Assess the Safety and Efficacy of Agents Targeting DNA Damage Repair in Combination With Olaparib Versus Olaparib Monotherapy in the Treatment of Metastatic Triple Negative Breast Cancer Patients Stratified by Alterations in Homologous Recombinant Repair (HRR)-Related Genes (Including BRCA1/2) (VIOLETTE).
Brief Title: To Assess Safety and Efficacy of Agents Targeting DNA Damage Repair With Olaparib Versus Olaparib Monotherapy.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5336C00001; 2017-002361-22 (EudraCT Number)
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Triple Negative Breast Cancer
Keywords: Germline BRCA mutation; Human epidermal growth factor receptor 2; Olaparib; Homologous Recombinant Repair (HRR)-related Genes
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ceralasertib; adavosertib; olaparib

STUDY DESIGN:
Masking Description: Given the study treatment design (monotherapy and 2 different combination therapies will be employed) neither patients nor Investigators will be blinded to study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Olaparib monotherapy (Active Comparator): All randomized patients will receive Olaparib monotherapy 300 mg twice daily (BD).
  Interventions: Drug: Olaparib Continuous (28-Day cycle) 300 mg BD.
- Olaparib+Ceralasertib (Active Comparator): All randomized patients will receive Olaparib 300 mg twice daily+Ceralasertib 160 mg once daily (OD).
  Interventions: Drug: Ceralasertib 160 mg OD + olaparib continuous 300 mg BD (28-day cycle).
- Olaparib+adavosertib (Active Comparator): All randomized patients will receive Olaparib 200 mg BD +adavosertib 150 mg BD. Following the discontinuation of adavosertib+olaparib treatment arm on 18 April 2019, patients receiving treatment with adavosertib+olaparib treatment were offered the opportunity to continue treatment on olaparib monotherapy at the approved dose (300 mg bd).
  Interventions: Drug: Adavosertib 150 mg BD + olaparib 200 mg BD (21-day cycle).

INTERVENTIONS:
Drug: Olaparib Continuous (28-Day cycle) 300 mg BD. — Two (2) 150 mg olaparib tablets should be taken at the same time each day, approximately 12 hours apart with one glass of water (approximately 250 mL).
  Arms: Olaparib monotherapy
Drug: Ceralasertib 160 mg OD + olaparib continuous 300 mg BD (28-day cycle). — Patients will be administered Ceralasertib OD at 160 mg from Day 1 to Day 7 (inclusive) of every 28-day cycle.
  Arms: Olaparib+Ceralasertib
Drug: Adavosertib 150 mg BD + olaparib 200 mg BD (21-day cycle). — Patients will be administered adavosertib BD at 150mg from Day 1 to Day 3 and Day 8 to Day 10.
  Arms: Olaparib+adavosertib

SUMMARY:
This study is to assess the efficacy and safety of olaparib monotherapy versus olaparib in combination with an inhibitor of ATR (Ataxia-Telangiectasia Mutated (ATM) and Rad3-related protein kinase (Ceralasertib [AZD6738]) and olaparib monotherapy versus olaparib in combination with an inhibitor of WEE1 (adavosertib [AZD1775]) in second or third line setting in patients with Triple-negative breast cancer (TNBC) prospectively stratified by presence/absence of qualifying tumour mutation in genes involved in the homologous recombination repair (HRR) pathway. Treatment arms are olaparib monotherapy, olaparib+ Ceralasertib and olaparib+adavosertib. The study subject population will be divided into Stratum A, Stratum B, and Stratum C. Due to the different schedules of administration of each of the treatment options as well as their different toxicity profiles, the study is not blinded. Study has two stage consent process- stage 1 consent (molecular screening for HRR defects) and stage 2 consent (main study). Patients with TNBC and with known qualifying BRCAm, non BRCAm HRRm and non HRRm status will be offered the option of consenting to the main part of the study within the 28-day screening period. Following the ISRC meeting on 17 April 2019 a recommendation was made to close the adavosertib+olaparib treatment arm across all biomarker strata. Patients receiving treatment with adavosertib+olaparib treatment were offered the opportunity to continue treatment on olaparib monotherapy at the approved dose (300 mg bd). Following the closure of this arm the total number of patients randomised will be lower (approximately 350 patients). Approximately 300 patients will be randomised (using randomisation ratio 1:1) to 2 ongoing treatment arms plus an additional 47 patients to a 3rd arm (olaparib+adavosertib) prior to the arm being discontinued.

DETAILED DESCRIPTION:
This is a prospective, open label, randomised, multi-centre Phase 2 study that will assess the efficacy and safety of olaparib monotherapy versus olaparib in combination with an inhibitor of ATR (Ceralasertib) and olaparib monotherapy versus olaparib in combination with an inhibitor of WEE1 (adavosertib) in second or third line setting in patients with TNBC prospectively stratified by presence/absence of qualifying tumour mutation in genes involved in the HRR pathway.

Eligible patients will be randomised by a ratio 1:1:1 to treatment Arm 1: olaparib continuous in a 28-day cycle, Arm 2: Ceralasertib Days 1-7 with olaparib continuous in a 28-day cycle or Arm 3: adavosertib Days 1-3 and 8-10 with olaparib continuous in a 21-day cycle. Following the ISRC meeting on 17 April 2019 a recommendation was made to close the adavosertib+olaparib treatment arm across all biomarker strata. Following closure of this arm the randomisation ratio will be 1:1 to olaparib monotherapy or Ceralasertib+olaparib. Patients who were receiving treatment with adavosertib+olaparib treatment were offered the opportunity to continue treatment on olaparib monotherapy at the approved dose (300 mg bd).

The study subject population will be divided into Stratum A (patients with mutations in BRCA1 or BRCA2 (Breast cancer susceptible gene mutation (BRCAm)), Stratum B (patients with mutations in any of the other genes involved in the HRR pathway and no mutation in BRCA1 and no mutation in BRCA2), and Stratum C (patients with no detected tumour mutations in any of the HRR genes). Within each stratum A, B and C, there will be further stratification by whether the patient received prior platinum-based therapy.

In the olaparib monotherapy treatment arm as well as in the Ceralasertib+olaparib treatment arm, patients will be administered olaparib bd at 300 mg continuously. Two (2) 150 mg olaparib tablets will be taken at the same time each day, approximately 12 hours apart with one glass of water (approximately 250 mL). In the adavosertib+olaparib treatment arm, patients will be given olaparib 200 mg bd (2 x 100 mg tablets twice a day) and adavosertib 150 mg bd from Day 1 to Day 3 (inclusive) and Day 8 to Day 10 (inclusive) of every 21-day cycle. Ceralasertib will be supplied as 20 mg, 80 mg, or 100 mg film coated tablets. Patients will be administered Ceralasertib od at 160 mg from Day 1 to Day 7 (inclusive) of every 28-day cycle. A total of 160 mg of Ceralasertib tablets will be taken at the same time on each day of dosing with approximately 250 mL of water. Adavosertib will be supplied as capsules containing 25 mg, 50 mg, 75 mg, 100 mg, or 200 mg of drug substance. Adavosertib will be taken with approximately 250 mL of water approximately 2 hours before or 2 hours after food. Olaparib, Ceralasertib and adavosertib will be provided by AstraZeneca.

Primary outcome measures (progression free survival [PFS]) will be analysed for the 3 patient populations BRCAm, Non BRCAm HRRm (Homologous Recombination Repair gene mutation) and Non HRRm. Secondary outcome measures will be analysed in 2 patient populations HRRm and All for PFS, Objective response rate (ORR) and overall survival (OS) will be analysed in all 5 patient populations. DoR, and tumour change will be analysed in BRCAm, Non BRCAm HRRm, and Non HRRm patient populations. Tumour and germline mutation status will be analysed only in the all patient population. PK outcome measures will be analysed only in the all patient population. Blinded Independent Central Review (BICR) of radiological imaging data will be carried out using RECIST version 1.1 and Investigator assessments will also be analysed for sensitivity purposes.

ELIGIBILITY:
Pertinent Inclusion criteria:

1. Informed consent prior to any study specific procedures.
2. Male or female ≥18 years of age.
3. Progressive cancer at the time of study entry.
4. Histologically or cytologically confirmed TNBC at initial diagnosis with evidence of metastatic disease and HER2 negative as per ASCO-CAP HER2 guideline recommendations 2013.
5. Patients must have received at least 1 and no more than 2 prior lines of treatment for metastatic disease with an anthracycline (eg, doxorubicin, epirubicin) and/or a taxane (eg, paclitaxel, docetaxel) unless contraindicated, in either the neo-adjuvant, adjuvant or metastatic setting.
6. Confirmed presence of qualifying HRR mutation or absence of any HRR mutation in tumour tissue by the Lynparza HRR assay.
7. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.
8. Patients must have normal organ and bone marrow function measured within 28 days prior to randomization (defined in the protocol).
9. ECOG PS 0-1 within 28 days of randomisation.
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential (contraception restrictions apply to participants and their partners).

13. Patient is willing to comply with the protocol requirements. 14. Life expectancy of ≥16 weeks.

Pertinent Exclusion criteria:

1. Cytotoxic chemotherapy, hormonal or non hormonal targeted therapy within 21 days of Cycle 1 Day 1 is not permitted. Palliative radiotherapy must have been completed 21 or more days before Cycle 1 Day 1. The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 5 days prior to study treatment.
2. More than 2 prior lines of cytotoxic chemotherapy for metastatic disease (prior treatments with hormonal, non-hormonal, biologics or the combination of an aromatase inhibitor and everolimus are not counted as a prior line of therapy).
3. Previous randomisation in the present study.
4. Previous treatment with a PARP inhibitor (including olaparib) or other DDR inhibitor (unless less than 3 weeks duration and at least 12 months has elapsed between the last dose and randomization).
5. Exposure to a small molecule IP within 30 days or 5 half-lives (whichever is longer) prior to randomisation. The minimum washout period for immunotherapy shall be 42 days.
6. Patients with second primary cancer (exceptions defined in the protocol).
7. Mean resting corrected QTc interval using the Fridericia formula (QTcF) >470 msec/female patients and >450 msec for male patients (as calculated per institutional standards) obtained from 3 ECGs performed 2-5 minutes apart at study entry, or congenital long QT syndrome.
8. Any of the following cardiac diseases currently or within the last 6 months: unstable angina pectoris, congestive heart failure ≥ Class 2 as defined by the New York Heart Association, acute myocardial infarction, conduction abnormality not controlled with pacemaker or medication (patients with a conduction abnormality controlled with pacemaker or medication at the time of screening are eligible), significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
9. Concomitant use of known strong or moderate cytochrome P (CYP) 3A inhibitors, strong or moderate CYP3A inducers, or sensitive CYP3A4 substrates or CYp3A4 substrates with a narrow therapeutic index (No longer applicable from CSPv7.0).
10. Persistent toxicities (≥ CTCAE grade 2) caused by previous cancer therapy, excluding alopecia and CTCAE grade 2 peripheral neuropathy.
11. Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
12. Immunocompromised patients, eg, human immunodeficiency virus (HIV).
13. Patients with known active hepatitis (ie, hepatitis B or C).
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non malignant systemic disease or active, uncontrolled infection.
15. Patients with symptomatic uncontrolled brain metastases.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
17. Patients with a known hypersensitivity to olaparib, adavosertib, Ceralasertib, or any of the excipients of the products.
18. Pregnant or breast feeding women.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2025-12-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tutt, MB ChB PhD, Principal Investigator — Guy's Hospital, Great Maze Pond, London.
Locations (124):
- United States (20):
  - Research Site, Birmingham, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Gilbert, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Chicago, Illinois
  - Research Site, Munster, Indiana
  - Research Site, Hazard, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Towson, Maryland
  - Research Site, Brick, New Jersey
  - Research Site, East Setauket, New York
  - Research Site, Lake Success, New York
  - Research Site, Mineola, New York
  - Research Site, Mount Kisco, New York
  - Research Site, Stony Brook, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Knoxville, Tennessee
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Belgium (8):
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Ottignies
  - Research Site, Wilrijk
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- Czechia (3):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- France (13):
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (7):
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Witten
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- Italy (19):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cona
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Macerata
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Siena
  - Research Site, Torino
- Netherlands (3):
  - Research Site, Breda
  - Research Site, Rotterdam
  - Research Site, The Hague
- Poland (10):
  - Research Site, Dąbrowa Górnicza
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Grzepnica
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (4):
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- South Korea (6):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (10):
  - Research Site, Barcelona
  - Research Site, Cáceres
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, San Sebastián
  - Research Site, Sant Cugat del Vallès
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Vigo
  - Research Site, Zaragoza
- Taiwan (5):
  - Research Site, Changhua
  - Research Site, Kaohsiung Hsien
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (10):
  - Research Site, Aberdeen
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Durham
  - Research Site, Edinburgh
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5336C00001&attachmentIdentifier=ec083208-5f73-415d-9a54-ba707ba58435&fileName=SAP_version_2.0_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5336C00001&attachmentIdentifier=9b2a32a3-1f1e-449b-8afa-319cc2e2a91e&fileName=Protocol_version_7.0_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5336C00001&attachmentIdentifier=49b53b42-fe19-4e60-aea7-829983b0ffe8&fileName=CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 21-Feb-2018 and 13-Nov-2020 in 15 countries in Asia, Europe, and North America.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the schedule of assessment.
Groups:
- Olaparib Monotherapy: Randomized patients received olaparib monotherapy 300 mg twice daily (BD) [28-day cycle], until objective radiological disease progression as per Response Evaluation Criteria In Solid Tumours Version (RECIST 1.1) as assessed by the Investigator or until any other discontinuation criteria were met.
- Olaparib + Ceralasertib: Randomized patients received ceralasertib 160 mg once daily (OD) from Days 1 to 7 and olaparib 300 mg twice daily (28-day cycle), until objective radiological disease progression as per RECIST 1.1 as assessed by the Investigator or until any other discontinuation criteria were met.
- Olaparib + Adavosertib: Randomized patients received adavosertib 150 mg BD from days 1 to 3 and days 8 to 10 and olaparib 200 mg BD (21-day cycle), until objective radiological disease progression as per RECIST 1.1 as assessed by the Investigator or until any other discontinuation criteria were met. The adavosertib dose was reduced from 175 mg to 150 mg BD through implementation of clinical study protocol (CSP) version 5.0.
Period: Overall Study
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Started | 114 | 112 | 47
Completed | 52 | 47 | 32
Not Completed | 62 | 65 | 15
Not completed — Patients ongoing study | 62 | 65 | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set: All randomized patients were analyzed according to the randomization scheme, regardless of the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib | Total
Number analyzed (Participants) | 114 | 112 | 47 | 273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.55) | 54.4 (10.85) | 52.7 (11.29) | 53.6 (11.21)
Age, Customized [Count of Participants; unit: Participants]
  <40 Years | 15 | 9 | 4 | 28
  >=40 to <50 Years | 30 | 27 | 18 | 75
  >=50 to <65 Years | 52 | 57 | 16 | 125
  >=65 to <75 Years | 14 | 13 | 8 | 35
  >=75 Years | 3 | 6 | 1 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 112 | 47 | 273
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 5 | 18
  Not Hispanic or Latino | 92 | 97 | 40 | 229
  Unknown or Not Reported | 16 | 8 | 2 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 23 | 7 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 81 | 77 | 34 | 192
  More than one race | 5 | 5 | 2 | 12
  Unknown or Not Reported | 12 | 7 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Per Stratum (BICR)
Description: Progression-free survival was defined as time from randomization until the date of objective disease progression or death, regardless of whether the patient withdrew from randomized therapy or received another anti-cancer therapy prior to progression. Progression was determined by Blinded independent central review (BICR) using Response Evaluation Criteria In Solid Tumours Version (RECIST 1.1). Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment. If patients had no evaluable visits or baseline data, the patient was censored at Study Day 1, unless death occurred within 17 weeks i.e., death within 17 weeks was relative to randomization. Here, the study patient population was stratified as follows: Breast cancer susceptible gene mutation (BRCAm) patients; non BRCAm homologous recombination repair gene mutation (HRRm) patients; non HRRm patients.
Time Frame: Until date of first documented progression or censoring date or date of death from any cause, whichever came first (assessed up to 32 months)
Population: All randomized patients were analyzed according to the randomisation scheme, regardless of the treatment they actually received. Here, number analyzed reflects number of patients enrolled in each stratum per treatment arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Months
  BRCAm patients: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients | 7.3 [5.5 to 8.1] | 7.4 [5.3 to 7.8] | 3.8 [3.7 to 11.4]
  non BRCAm HRRm patients: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm patients | 1.9 [1.8 to 3.6] | 3.9 [1.9 to 17.4] | 2.1 [0.6 to 14.1]
  non HRRm patients: number analyzed (Participants) | 51 | 52 | 27
  non HRRm patients | 1.9 [1.8 to 2.9] | 3.6 [2.7 to 3.8] | 4.4 [3.2 to 5.6]
Statistical Analysis 1: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population BRCAm; Test type: Superiority; p = 0.9403, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 1.02, 90% CI 2-sided [0.63 to 1.66] — Proportional hazards models based on prior platinum-based therapy (no, yes). Hazard ratio < 1 favours respective combination treatment related with a longer PFS than olaparib monotherapy. Here, favours olaparib monotherapy
Statistical Analysis 2: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population BRCAm; Test type: Superiority; p = 0.9282, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 1.01, 90% CI 2-sided [0.52 to 1.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population Non BRCAm HRRm; Test type: Superiority; p = 0.1274, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.54, 90% CI 2-sided [0.28 to 1.03] — Proportional hazards models based on prior platinum-based therapy (no, yes). Hazard ratio < 1 favours respective combination treatment related with a longer PFS than olaparib monotherapy. Here, favours olaparib + ceralasertib
Statistical Analysis 4: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population Non BRCAm HRRm; Test type: Superiority; p = 0.2956, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.56, 90% CI 2-sided [0.23 to 1.26] — Proportional hazards models based on prior platinum-based therapy (no, yes). Hazard ratio < 1 favours respective combination treatment related with a longer PFS than olaparib monotherapy. Here, favours olaparib + adavosertib
Statistical Analysis 5: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population Non HRRm; Test type: Superiority; p = 0.2959, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.76, 90% CI 2-sided [0.50 to 1.14] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 6: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population Non HRRm; Test type: Superiority; p = 0.0193, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.48, 90% CI 2-sided [0.28 to 0.80] — [estimate comment as in outcome 1, analysis 4]

2. Primary Outcome: Progression-free Survival Per Stratum (Sensitivity Analysis)
Description: Progression-free survival was defined as time from randomization until the date of objective disease progression or death, regardless of whether the patient withdrew from randomized therapy or received another anti-cancer therapy prior to progression. Progression was determined by the site Investigator. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment. If patients had no evaluable visits or baseline data, the patient was censored at Study Day 1, unless death occurred within 17 weeks i.e., death within 17 weeks was relative to randomization. Here, the study patient population was stratified as follows: BRCAm patients; non BRCAm HRRm patients; non HRRm patients.
Time Frame: as for outcome 1
Population: All randomized patients were analyzed according to the randomisation scheme, regardless of the treatment actually they received. Here, number analyzed reflects number of patients enrolled in each stratum per treatment arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Months
  BRCAm patients: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients | 7.4 [5.6 to 10.0] | 7.5 [5.7 to 9.3] | 5.4 [3.7 to 11.5]
  non BRCAm HRRm patients: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm patients | 3.4 [1.8 to 3.7] | 3.7 [1.9 to 5.5] | 2.9 [1.0 to 7.4]
  non HRRm patients: number analyzed (Participants) | 51 | 52 | 27
  non HRRm patients | 1.9 [1.7 to 2.4] | 3.5 [1.9 to 3.8] | 2.9 [1.9 to 4.0]
Statistical Analysis 1: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population BRCAm; Test type: Superiority; p = 0.6147, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.87, 90% CI 2-sided [0.53 to 1.39] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 2: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population BRCAm; Test type: Superiority; p = 0.7879, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.93, 90% CI 2-sided [0.48 to 1.68] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 3: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population Non BRCAm HRRm; Test type: Superiority; p = 0.3695, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.71, 90% CI 2-sided [0.38 to 1.31] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population Non BRCAm HRRm; Test type: Superiority; p = 0.4586, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.71, 90% CI 2-sided [0.29 to 1.58] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Olaparib Monotherapy vs Olaparib + Ceralasertib; Patient Population Non HRRm; Test type: Superiority; p = 0.7452, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.89, 90% CI 2-sided [0.61 to 1.31] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 6: Comparison: Olaparib Monotherapy vs Olaparib + Adavosertib; Patient Population Non HRRm; Test type: Superiority; p = 0.1185, Two-sided log-rank tests; Stratified for prior platinum-based therapy (no,yes) using Breslow's approach for handling of ties; Hazard Ratio (HR) = 0.61, 90% CI 2-sided [0.37 to 1.00] — [estimate comment as in outcome 1, analysis 4]

3. Secondary Outcome: Progression-free Survival (Per BICR)
Description: Progression-free survival was defined as time from randomization until the date of objective disease progression or death, regardless of whether the patient withdrew from randomized therapy or received another anti-cancer therapy prior to progression. Progression was determined by BICR using RECIST 1.1. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment. If patients had no evaluable visits or baseline data, the patient was censored at Study Day 1, unless death occurred within 17 weeks i.e., death within 17 weeks was relative to randomization. Here, the study patient population was presented as follows: HRRm and all enrolled patients.
Time Frame: From randomization until date of first documented progression or censoring date or date of death from any cause, whichever came first (assessed up to 32 months)
Population: All randomized patients were analyzed according to the randomization scheme, regardless of the treatment they actually received. Here, number analyzed reflects number of patients enrolled in each stratum per treatment arm.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Months
  HRRm patients per BICR: number analyzed (Participants) | 63 | 60 | 20
  HRRm patients per BICR | 5.6 [3.7 to 6.1] | 5.6 [5.3 to 7.4] | 3.7 [3.4 to 7.4]
  All patients per BICR | 3.6 [2.9 to 5.4] | 5.3 [3.7 to 5.5] | 3.8 [3.7 to 5.6]

4. Secondary Outcome: Number of Patients With Objective Response (Per BICR and Per Sensitivity Analysis)
Description: The objective response was defined as patients with at least one BICR assessed visit response of CR or PR. For sensitivity analysis, objective response was defined as the patients with at least one visit response of CR or PR based on Investigator data. These are unadjusted percentages of responders (100 * number of responders / number of patients in full analysis set). The objective response was assessed per RECIST 1.1 guidelines for: measurable lesions (measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) using CT or MRI, non-measurable lesions (all other lesions, including small lesions (longest diameter <10 mm or pathological lymph nodes with ≥10 to <15mm short axis at baseline), based on target lesions [TL] (maximum of 5 measurable lesions (with a maximum of 2 lesions per organ), non-target lesions [NTL] (lesions (or sites of disease) not recorded as TL should be identified as NTL at baseline) and any new lesions.
Time Frame: From date of randomization until date of first documented progression or last evaluable assessment, or start of subsequent anti-cancer therapy (Whichever occurred first [assessed up to 32 months])
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Participants
  BRCAm patients per BICR: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients per BICR | 19 | 20 | 6
  non BRCAm HRRm patients per BICR: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm patients per BICR | 3 | 4 | 0
  non HRRm patients per BICR: number analyzed (Participants) | 51 | 52 | 27
  non HRRm patients per BICR | 2 | 8 | 3
  HRRm patients per BICR: number analyzed (Participants) | 63 | 60 | 20
  HRRm patients per BICR | 22 | 24 | 6
  All patients per BICR | 24 | 32 | 9
  BRCAm patients per sensitivity analysis: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients per sensitivity analysis | 18 | 20 | 7
  non BRCAm HRRm per sensitivity analysis: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm per sensitivity analysis | 3 | 4 | 1
  non HRRm per sensitivity analysis: number analyzed (Participants) | 51 | 52 | 27
  non HRRm per sensitivity analysis | 1 | 11 | 3

5. Secondary Outcome: Objective Response Rate (ORR) (Per BICR and Per Sensitivity Analysis)
Description: The ORR was defined using BICR data to define a visit response of CR or PR, with denominator defined as number of patients in FAS. For sensitivity analysis, ORR is defined as the percentage of patients with at least one investigator-assessed visit response of CR or PR, with denominator defined as number of patients in FAS. These are summarized using adjusted response rates, which are computed with a logistic regression including factors study treatment and prior platinum-based therapy (no, yes), i.e. these response rates are adjusted for prior platinum-based therapy, which is one of the randomisation stratification factors. The adjusted response rates have been presented as a percentage of patients.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Number; unit: Percentage of patients
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Percentage of patients
  BRCAm patients per BICR: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients per BICR | 42.7 | 48.4 | 44.9
  non BRCAm HRRm patients per BICR: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm patients per BICR | 15.0 | 20.0 | 0.0
  non HRRm patients per BICR: number analyzed (Participants) | 51 | 52 | 27
  non HRRm patients per BICR | 3.9 | 15.4 | 11.1
  HRRm patients per BICR: number analyzed (Participants) | 63 | 60 | 20
  HRRm patients per BICR | 33.2 | 38.0 | 28.5
  All patients per BICR | 20.1 | 27.3 | 18.3
  BRCAm patients per sensitivity analysis: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients per sensitivity analysis | 41.0 | 49.0 | 53.1
  non BRCAm HRRm per sensitivity analysis: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm per sensitivity analysis | 15.0 | 20.0 | 14.3
  non HRRm per sensitivity analysis: number analyzed (Participants) | 51 | 52 | 27
  non HRRm per sensitivity analysis | 2.0 | 21.2 | 11.1

6. Secondary Outcome: Duration of Response (DoR) [Per BICR and Per Sensitivity Analysis]
Description: The DoR was defined as the time from the date of first documented response according to BICR data until date of documented progression according to BICR data or death in the absence of disease progression. For sensitivity analysis, DoR was defined as the time from the date of first documented response according to Investigator assessment until date of documented progression according to Investigator assessment or death in the absence of disease progression. Here, the median DoR and the 25th and 75th percentile of DoR are presented. The DoR from onset of response was calculated using Kaplan-Meier technique. Here, the study patient population was stratified as follows: BRCAm patients; non BRCAm HRRm patients; non HRRm patients.
Time Frame: From date of first documented response until date of first documented progression or last evaluable assessment (assessed up to 32 months)
Population: All randomized patients were analyzed according to the randomization scheme, regardless of the treatment they actually received. Here, number analyzed reflects number of patients with objective response.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Weeks
  BRCAm patients per BICR: number analyzed (Participants) | 19 | 20 | 6
  BRCAm patients per BICR | 20.0 [16.0 to 32.1] | 32.0 [16.1 to 56.4] | 33.4 [8.1 to 42.1]
  non BRCAm HRRm patients per BICR: number analyzed (Participants) | 3 | 4 | 0
  non BRCAm HRRm patients per BICR | 16.8 [16.3 to 17.3] | 17.1 [12.3 to NA] — Not calculable due to insufficient follow-up |
  non HRRm patients per BICR: number analyzed (Participants) | 2 | 8 | 3
  non HRRm patients per BICR | 11.4 [7.1 to 15.7] | 24.1 [15.1 to 24.1] | 16.6 [16.1 to 17.0]
  BRCAm patients per sensitivity analysis: number analyzed (Participants) | 18 | 20 | 7
  BRCAm patients per sensitivity analysis | 20.0 [15.1 to 42.6] | 32.6 [24.1 to 93.4] | 41.1 [16.1 to NA] — Not calculable due to insufficient follow-up
  non BRCAm HRRm per sensitivity analysis: number analyzed (Participants) | 3 | 4 | 1
  non BRCAm HRRm per sensitivity analysis | 16.3 [8.1 to 28.1] | 16.5 [12.0 to 17.1] | 48.1 [48.1 to 48.1]
  non HRRm per sensitivity analysis: number analyzed (Participants) | 1 | 11 | 3
  non HRRm per sensitivity analysis | 13.6 [13.6 to 13.6] | 11.7 [8.1 to 16.1] | 31.6 [31.3 to 31.9]

7. Secondary Outcome: Percentage Change From Baseline in Target Lesion Tumour Size [Per BICR and Per Sensitivity Analysis]
Description: Tumour size was the sum of the longest diameters of the target lesions (TLs). The percentage change in TL tumour size at Week 16 was obtained for each patient as follows (considering a visit window around the scheduled day of the Week 16 assessment): (TL at Week 16 minus TL at baseline) divided by (TL at baseline) multiplied by 100. Here, the percentage change data have been reported as per BICR and as per sensitivity analysis per investigator assessments. Here, the study patient population was stratified as follows: BRCAm patients; non BRCAm HRRm patients; non HRRm patients.
Time Frame: Baseline, at Week 16
Population: All randomized patients were analyzed according to the randomization scheme, regardless of the treatment they actually received. Here, number analyzed reflects the number of patients with an observed or imputed value for the percentage change from baseline at week 16.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Percentage change
  BRCAm patients per BICR: number analyzed (Participants) | 32 | 34 | 11
  BRCAm patients per BICR | -27.7 (34.33) | -33.8 (37.77) | -34.1 (42.52)
  non BRCAm HRRm patients per BICR: number analyzed (Participants) | 18 | 18 | 5
  non BRCAm HRRm patients per BICR | 4.9 (35.78) | 4.9 (35.72) | 42.3 (27.44)
  non HRRm patients per BICR: number analyzed (Participants) | 45 | 46 | 20
  non HRRm patients per BICR | 40.3 (76.18) | 5.7 (40.46) | 9.2 (32.66)
  BRCAm patients per sensitivity analysis: number analyzed (Participants) | 35 | 36 | 12
  BRCAm patients per sensitivity analysis | -21.9 (39.88) | -29.5 (35.36) | -23.7 (41.85)
  non BRCAm HRRm per sensitivity analysis: number analyzed (Participants) | 18 | 19 | 7
  non BRCAm HRRm per sensitivity analysis | 6.2 (34.77) | -2.1 (40.66) | 73.9 (107.94)
  non HRRm per sensitivity analysis: number analyzed (Participants) | 48 | 51 | 23
  non HRRm per sensitivity analysis | 20.1 (34.71) | 3.9 (37.20) | 9.3 (27.46)

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomisation until death due to any cause. Any patient not known to have died at the time of data cut-off was censored based on the last recorded date on which the patient was known to be alive. Here, the study patient population was stratified as follows: BRCAm patients; non BRCAm HRRm patients; non HRRm patients.
Time Frame: From the date of randomisation until time of data cut-off date or death due to any cause (assessed up to 32 months)
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 114 | 112 | 47
Months
  BRCAm patients: number analyzed (Participants) | 43 | 40 | 13
  BRCAm patients | 20.4 [16.1 to 22.0] | 15.5 [13.0 to NA] — Not calculable due to insufficient follow-up | 22.8 [12.1 to NA] — Not calculable due to insufficient follow-up
  non BRCAm HRRm patients: number analyzed (Participants) | 20 | 20 | 7
  non BRCAm HRRm patients | 8.4 [6.2 to 14.1] | 12.4 [7.9 to NA] — Not calculable due to insufficient follow-up | 8.0 [1.0 to NA] — Not calculable due to insufficient follow-up
  non HRRm patients: number analyzed (Participants) | 51 | 52 | 27
  non HRRm patients | 9.2 [6.9 to NA] — Not calculable due to insufficient follow-up | 10.3 [7.3 to NA] — Not calculable due to insufficient follow-up | 10.6 [7.2 to 14.2]

9. Secondary Outcome: Plasma Drug Concentrations of Olaparib
Description: Plasma drug concentrations of olaparib are evaluated to assess exposure to olaparib in all patients.
Time Frame: Pre-dose at Cycle 1 Day 7 [olaparib monotherapy or ceralasertib+olaparib] or Cycle 1 Day 10 [adavosertib+olaparib] (each cycle is 21 days for olaparib+adavosertib, and 28 days for olaparib monotherapy and olaparib+ceralasertib)
Population: Pharmacokinetic (PK) analysis set included patients who have received at least one dose of study medication per the protocol and for whom there was at least one reportable PK concentration.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 94 | 85 | 36
ug/mL | 2.97 (2.41) | 2.90 (2.68) | 3.22 (3.37)

10. Secondary Outcome: Plasma Drug Concentrations of Ceralasertib and Adavosertib
Description: Plasma drug concentrations of ceralasertib and adavosertib are evaluated to assess exposure to ceralasertib and adavosertib in all patients.
Time Frame: Pre-dose at Cycle 1 Day 7 [ceralasertib+olaparib] or Cycle 1 Day 10 [adavosertib+olaparib] (each cycle is 21 days for olaparib+adavosertib, and 28 days for olaparib+ceralasertib)
Population: PK analysis set included patients who have received at least one dose of study medication per the protocol and for whom there was at least one reportable PK concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 89 | 39
ng/mL | 870.05 (772.05) | 290.46 (169.07)

11. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events reported after treatment with olaparib monotherapy, the combination of ceralasertib and olaparib or the combination of adavosertib and olaparib. The data includes adverse events (AEs) with an onset or worsening date on or after the date of first dose and up to and including 30 days following the date of last dose of study medication.
Time Frame: From screening until Follow-up 30 Days after last dose of study treatment (assessed up to 32 months)
Population: The safety analysis set included all patients who received at least one dose of randomized treatment according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
Number analyzed (Participants) | 110 | 109 | 46
Participants
  Any AE | 105 | 107 | 46
  Any AE causally related to olaparib | 91 | 95 | 43
  Any AE causally related to non-olaparib | NA — In this arm patients have received only olaparib | 92 | 45
  Any AE causally related to non-olaparib and olaparib | NA — In this arm patients have received only olaparib | 91 | 42
  Any AE with outcome = death | 1 | 2 | 1
  Any AE with outcome = death, causally related to olaparib | 0 | 0 | 0
  Any AE with outcome = death, causally related to non-olaparib | NA — In this arm patients have received only olaparib | 0 | 0
  Any AE with outcome = death, causally related to non-olaparib and olaparib | NA — In this arm patients have received only olaparib | 0 | 0
  Any SAE | 21 | 24 | 17
  Any SAE causally related to olaparib | 4 | 9 | 9
  Any SAE causally related to non-olaparib | NA — In this arm patients have received only olaparib | 7 | 14
  Any SAE causally related to non-olaparib and olaparib | NA — In this arm patients have received only olaparib | 7 | 9
  Any AE leading to discontinuation of study treatment | 2 | 12 | 9
  AEs leading to reduction of study treatment | 15 | 32 | 19
  AEs leading to reduction of olaparib | 15 | 30 | 11
  AEs leading to reduction of non-olaparib | NA — In this arm patients have received only olaparib | 16 | 12
  AEs leading to reduction of non-olaparib and olaparib | NA — In this arm patients have received only olaparib | 11 | 3

ADVERSE EVENTS:
Time Frame: From screening until Follow-up 30 Days after last dose of study treatment (assessed up to 32 months)
Description: Full analysis set population is used for All-cause Mortality as death formed part of efficacy. However, safety analysis set is used for serious adverse events and non-serious adverse event as the adverse events form part of safety and not efficacy.
Arm/Group | Olaparib Monotherapy | Olaparib + Ceralasertib | Olaparib + Adavosertib
All-Cause Mortality (participants affected / at risk) | 42/114 | 40/112 | 26/47
Serious Adverse Events (participants affected / at risk) | 21/110 | 24/109 | 17/46
Other Adverse Events (participants affected / at risk) | 99/110 | 106/109 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib Monotherapy (N=110) | Olaparib + Ceralasertib (N=109) | Olaparib + Adavosertib (N=46)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib Monotherapy (N=110) | Olaparib + Ceralasertib (N=109) | Olaparib + Adavosertib (N=46)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 36 (51) | 56 (99) | 23 (45)
Leukopenia (Blood and lymphatic system disorders) | 5 (7) | 7 (12) | 8 (15)
Neutropenia (Blood and lymphatic system disorders) | 10 (18) | 20 (29) | 19 (39)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 12 (16) | 9 (23)
Decreased appetite (Metabolism and nutrition disorders) | 19 (23) | 22 (22) | 10 (13)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5)
Dizziness (Nervous system disorders) | 8 (9) | 11 (12) | 3 (7)
Headache (Nervous system disorders) | 13 (19) | 16 (18) | 4 (7)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2) | 3 (5)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3) | 4 (4)
Hot flush (Vascular disorders) | 0 (0) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 5 (9) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 10 (11) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 11 (12) | 8 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 7 (10) | 6 (9)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 7 (8) | 2 (3)
Constipation (Gastrointestinal disorders) | 12 (15) | 17 (19) | 10 (13)
Diarrhoea (Gastrointestinal disorders) | 16 (20) | 24 (44) | 25 (59)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 6 (6) | 3 (4)
Nausea (Gastrointestinal disorders) | 55 (75) | 64 (102) | 26 (42)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 8 (9) | 2 (2)
Vomiting (Gastrointestinal disorders) | 34 (49) | 31 (49) | 15 (32)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 9 (12) | 6 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 9 (11) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 3 (3)
Asthenia (General disorders) | 26 (34) | 33 (41) | 7 (10)
Fatigue (General disorders) | 30 (36) | 32 (52) | 16 (26)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 4 (4) | 6 (6) | 3 (3)
Pyrexia (General disorders) | 6 (6) | 7 (10) | 6 (7)
Alanine aminotransferase increased (Investigations) | 8 (9) | 7 (8) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 5 (6) | 7 (7)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (2) | 4 (6)
C-reactive protein increased (Investigations) | 3 (3) | 4 (4) | 4 (4)
Lymphocyte count decreased (Investigations) | 5 (5) | 3 (4) | 3 (4)
Neutrophil count decreased (Investigations) | 5 (6) | 8 (17) | 6 (12)
Platelet count decreased (Investigations) | 2 (6) | 10 (19) | 8 (16)
Weight decreased (Investigations) | 3 (3) | 3 (4) | 5 (5)
White blood cell count decreased (Investigations) | 3 (3) | 9 (15) | 8 (10)

LIMITATIONS AND CAVEATS:
The interpretation of efficacy results of the adavosertib + olaparib arm and comparison with the olaparib monotherapy arm and ceralasertib + olaparib arm is limited due to the lower number of patients with available data in the adavosertib + olaparib arm, the nature of the analysis (intent-to-treat), and the fact that some of the patients switched from adavosertib + olaparib treatment to olaparib monotherapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03330847/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT03330847/SAP_001.pdf